CLINICAL TRIAL: NCT07377760
Title: Adaptive Text Messaging Reminders Combined With Non-monetary Incentives to Improve Adherence to Antiretroviral Treatment Among Adolescents Living With HIV in Ethiopia: a Hybrid Effectiveness-implementation Trial
Brief Title: Adaptive Text Messaging and Non-Monetary Incentives to Sustain ART Adherence Among Adolescents Living With HIV in Ethiopia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arba Minch University (Other)
Responsible Party: Principal Investigator, Abayneh Tunje Tanga, Adaptive text messaging reminders combined with non-monetary incentives to improve adherence to antiretroviral treatment among adolescents in Ethiopia: a hybrid effectiveness-implementation trial, Arba Minch University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIPHER Research Grant IAS_146
Record Dates: First submitted 2026-01-01; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Antiretroviral Therapy (ART) Adherence Among Adolescents Living With HIV
Keywords: Adolescents with HIV; ART adherence; SMS reminders; habit-based digital intervention; cue-reward system; viral suppression; Ethiopia

STUDY DESIGN:
Intervention Model Description: Adolescents living with HIV are randomly assigned to two SMS-based habit-reward interventions or a standard care control group to evaluate ART adherence, retention, and health outcomes.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-adaptive reminder text messaging combined with non-monetary incentives (Experimental)
  Interventions: Behavioral: Adaptive interventions; Behavioral: The control arm
- Adaptive text messaging (Experimental)
  Interventions: Behavioral: Non-adaptive reminder text messaging; Behavioral: The control arm
- Control (standard care) (No Intervention)

INTERVENTIONS:
Behavioral: Non-adaptive reminder text messaging — Non-adaptive reminder text messaging combined with non-monetary incentives versus the standard of care. Under this sub-aim, we will compare adherence levels between those who receive continuous text messaging combined with participant-preferences of daily cue and medication time.
  Arms: Adaptive text messaging
Behavioral: Adaptive interventions — Participants will choose a lifestyle 'cue,' as in arm 1, and receive daily, personalized text message reminders tailored to their selected cues for the first three months. After three months, adherence will be evaluated, and a non-monetary reward will be provided to both adherent and non-adherent participants. Following this, the cue reminder text messages will be discontinued for participants who achieved 95% ART adherence over the next 12-month period. However, they will receive a non-monetary reward for achieving 95% ART adherence over six months of follow-up.
  Arms: Non-adaptive reminder text messaging combined with non-monetary incentives
Behavioral: The control arm — In the control arm, all adolescents will receive the standard care as per the national guidelines (25). The standard care provided encompasses counseling, mental health support, nutritional assessment, and social and emotional support given by family, friends, and healthcare providers to adolescents diagnosed with HIV.
  Arms: Adaptive text messaging; Non-adaptive reminder text messaging combined with non-monetary incentives

SUMMARY:
Many adolescents living with HIV have difficulty taking their medicine on time, which can make it less effective and affect their health. This study will test whether sending reminder text messages, combined with small rewards like school supplies, hygiene kits, or sports items, can help adolescents take their HIV medicine regularly and stay in care. Each adolescent will choose a daily habit or routine to link to their medication. We will compare two groups receiving messages and rewards to a group receiving standard care to see which approach works best. We will also ask participants about their experience with the messages and rewards. The aim is to find a simple and effective way to help adolescents living with HIV stay healthy and in care.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adolescents aged 15 to 19 who have been on ART for at least a year and want to continue treatment at the selected facility during the trial period are eligible.

Exclusion Criteria:

* Participants outside of the specified age range.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 327 (Estimated)
Dates: Start 2026-03-09 (Estimated); Primary Completion 2027-03-12 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Adaptive text messaging reminders combined with non-monetary incentives to improve sustained adherence to antiretroviral treatment among adolescents in Ethiopia: a hybrid effectiveness-implementation trial | 12 months
  ART adherence will be measured using a multi-method composite adherence assessment tool based on previously validated measures, including self-reported adherence, pill count (PC), and retention in care (missed appointments). Self-reported adherence will be assessed through four validated yes/no questions addressing difficulties remembering medication, intentional discontinuation when feeling better or worse, and missed doses over the preceding four days. Participants will also rate their adherence over the past 30 days using a visual analogue scale (VAS) ranging from 0 (no adherence) to 10 (perfect adherence). Each adherence component will be dichotomized using established thresholds (≥95% adherence for self-report, pill count, and VAS; no missed appointments for retention in care) and assigned a score of 1 (adherent) or 0 (non-adherent). Component scores will be summed to generate a composite adherence index ranging from 0 to 3, which will be reported as a single adherence measure ca

SECONDARY OUTCOMES:
Implementation Outcomes of Adaptive SMS Reminders with Incentives for Adolescents Living with HIV | 3-12 months
  Implementation Outcomes: The delivery, uptake, and integration of the adaptive SMS reminder and non-monetary incentive intervention will be evaluated by assessing six key implementation outcomes: acceptability, feasibility, fidelity, adoption/uptake, penetration/reach, and sustainability/maintenance.
  Description of Outcome Measures:
  Acceptability: Measured using the validated Acceptability of Intervention Measure (AIM) and supplemented with in-depth qualitative interviews with participants regarding the intervention's content, timing, and incentives. Assessment timepoints: 3, 6, 9, and 12 months.
  Feasibility: Evaluated through digital logs of SMS delivery, records of incentive distribution, and semi-structured interviews with clinic staff to identify barriers, facilitators, and ease of implementation. Formally assessed at 6 and 12 months, with continuous process monitoring.
  Fidelity: Assessed by comparing the planned intervention protocol
Effect of Adaptive SMS and Incentives on 12-Month Viral Suppression in Adolescents with HIV | 12 months
  The proportion of adolescents living with HIV who maintain a viral load below 1,000 copies/mL at the 12-month study visit, assessed as the primary clinical effectiveness outcome of the adaptive SMS and incentive intervention
Cost-Effectiveness and Cost-Utility of Adaptive SMS Reminders with Non-Monetary Incentives for Improving ART Adherence Among Adolescents with HIV | 12 months
  This study will perform a comprehensive economic evaluation from both healthcare system and societal perspectives. The analysis will compare the incremental costs and health outcomes of the combined adaptive SMS reminder and non-monetary incentive intervention against the standard of care. Cost-effectiveness will be assessed as the incremental cost per additional adolescent achieving sustained ART adherence. Cost-utility will be measured as the incremental cost per Quality-Adjusted Life Year (QALY) gained, with health utilities derived from the EQ-5D-Y/3L instrument administered at baseline, 6, and 12 months. We will calculate Incremental Cost-Effectiveness Ratios (ICERs) and conduct sensitivity analyses to assess uncertainty. A budget impact analysis will model the financial consequences of potential scale-up.

OTHER OUTCOMES:
Patient-Level Psychosocial and Behavioral Determinants of ART Adherence | Measurement Time Points: Baseline, 3, 6, 9, and 12 months post-enrollment.
  This study will measure a comprehensive set of patient-level factors hypothesized to influence sustained adherence to antiretroviral therapy (ART) among adolescents living with HIV. Validated self-report scales will be used to assess habit strength, intrinsic motivation, HIV-related stigma, depressive symptoms, and perceived social support.
  Rationale for Measurement Schedule:
  Baseline: To establish initial levels, identify baseline predictors of subsequent adherence and viral load suppression/rebound, and allow for statistical adjustment of participant differences.
  3-Month Follow-up: To detect initial changes in psychosocial factors and investigate early mediators of adherence behavior following intervention initiation.
  6-Month Follow-up (Midline): To track short-term trends and identify adaptation or emerging challenges in adherence behavior.
  9- and 12-Month Follow-ups: To assess the longer-term trajector
Patient-Level Determinants and Contextual Factors | From baseline to 12-months
  Patient-level determinants, including habit strength, intrinsic motivation, HIV-related stigma, depressive symptoms, and social support, will be measured using validated self-report scales at baseline, 3, 6, 9, and 12 months. Baseline: Establish initial levels, identify predictors of adherence and viral suppression and its rebound, and allow adjustment for participant differences. Early follow-up (3 months): Detect initial changes and early mediators of adherence. Midline (6 months): Track short-term trends, adaptation, and challenges in adherence behavior. Later follow-ups (9 and 12 months): Assess longer-term changes and maintenance of psychosocial factors. These measures will be analyzed as potential mediators or moderators of sustained ART adherence and viral load suppression.

CONTACTS AND LOCATIONS:
Overall Officials: Degu J Dare, MD,PhD, Study Director — KNCV
Locations (1):
- Arba Minch University, Arba Minch, Ethiopia

REFERENCES:
- [Result] Hernell O, Egelrud T, Olivecrona T. Serum-stimulated lipases (lipoprotein lipases). Immunological crossreaction between the bovine and the human enzymes. Biochim Biophys Acta. 1975 Feb 13;381(2):233-41. PMID 46150
- [Result] Nachega JB, Mills EJ, Schechter M. Antiretroviral therapy adherence and retention in care in middle-income and low-income countries: current status of knowledge and research priorities. Curr Opin HIV AIDS. 2010;5(1):70-7.
- See also: Related Info — https://journals.lww.com/co-hivandaids/abstract/2010/01000/antiretroviral_therapy_adherence_and_retention_in.11.aspx